CLINICAL TRIAL: NCT04296058
Title: SOX4 Activates CXCL12 in Hepatocellular Carcinoma Cells to Modulate Endothelial Cell Migration and Angiogenesis in Vivo
Brief Title: The Mechanism of Sox4 Transcription in Regulation of Angiogenesis in Hepatocellular Carcinoma
Acronym: SOX4 in HCC
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 106-2314-B-182A-113; 103-2314-B-182A-082-MY1-3 (Other Grant/Funding Number: MOST); 106-2314-B-182A-113 (Other Grant/Funding Number: MOST); CMRPD1G0611 (Other Grant/Funding Number: Chang Gung medical foundation); CMRPD1H0661 (Other Grant/Funding Number: Chang Gung medical foundation); CMRPG1J0061 (Other Grant/Funding Number: Chang Gung medical foundation)
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2019-03

CONDITIONS: Translational Research of SOX4 in Hepatocellular Carcinoma
Keywords: SOX4; angiogenesis; microvessel density
MeSH Terms: interventions — Microvascular Density

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- SOX4 high: Nuclear expression of SOX4 over 90% in tumor specimen was defined as SOX4 high group
  Interventions: Other: microvessel density
- SOX4 low: Nuclear expression of SOX4 less than 90% in tumor specimen was defined as SOX4 low group
  Interventions: Other: microvessel density

INTERVENTIONS:
Other: microvessel density — the vessel numbers in high power field with Anti-CD31 staining in tumor specimen

SUMMARY:
Two hundred HCC patients with partial hepatectomy were enrolled as a cohort for observational study. The inclusion criterion was intended curative hepatectomy for HCC patients by image analysis, and the exclusion criteria were unresectable disease, synchronous cancers, recurrent cancers, or distant metastasis. The study endpoint was 30 March 2019, and tumor staging was based on the 8th edition of the American Joint Committee on Cancer (AJCC) TNM staging system for HCC

DETAILED DESCRIPTION:
To determine the role of SOX4 in tumor progression in patients with HCC, we examined SOX4 expression through immunohistochemistry (IHC) staining of 200 formalin-fixed and paraffin-embedded (FFPE) HCC specimens . The SOX4 high group of patients was associated with positive etiology of hepatitis B virus (P = 0.044), tumor size >5 cm (P = 0.014), thrombus formation (P = 0.012), higher microvessel density (MVD) (P = 0.012) in tumor lesions, and distant metastasis (P <0.001).

Cox regression analysis showed that patients with elderly age (P <0.001), higher ⍺-fetal protein (AFP) (P = 0.045), presence of cirrhosis (P = 0.008), and SOX4 high in tumor specimen (P = 0.042) were independent risk factors . The SOX4 high group performed significantly worse regarding overall survival (OS) (P = 0.043) and disease-free survival (DFS) (P = 0.019) based on the Kaplan-Meier analysis.

ELIGIBILITY:
Inclusion Criteria:

subjects with pathologic diagnosis of hepatocellular carcinoma and curative partial hepatectomies -

Exclusion Criteria:

history of different malignant disease, subject cannot be treated with curative surgery -

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects with pathologic diagnosis of hepatocellular carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-01-08 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Disease free survival (DFS) | a month
  The length of time from curative hepatectomies and recurrence or mortality

SECONDARY OUTCOMES:
Overall survival | a month
  The length of time from curative hepatectomies and still alive

IPD SHARING:
Plan to Share IPD: No